CLINICAL TRIAL: NCT01076881
Title: Combined Resistance and Aerobic Exercise is Better Than Resistance Training Alone to Improve Functional Performance of Hemodialysis Patients - Results of a Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Católica de Pelotas (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UCPelotas01
Record Dates: First submitted 2010-02-17; First posted 2010-02-26 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- combined aerobic and resistance training (Experimental)
  Interventions: Behavioral: exercise training
- resistance training alone (Active Comparator)
  Interventions: Behavioral: exercise training

INTERVENTIONS:
Behavioral: exercise training

SUMMARY:
This is a randomized trial with participants recruited from one dialysis unit of a Brazilian university hospital. Hemodialysis patients were assigned to receive the resistance exercise combined with an aerobic training or the resistance training alone for a period of 10 weeks. The functional performance of patients was assessed before and after the intervention through the six-minute walk test (6MWT). The difference over time of the 6MWT was compared between the groups through multivariate linear regression.

Thirteen patients were allocated for each group of intervention. The difference in distance walked before and after intervention in the combined training group was of +39.7 (61.4) meters, and this difference in the resistance training group was of -19.2 (53.9) meters, p=0.01. In multivariate analysis with adjustment for age, skin color, gender, hematocrit, time since starting dialysis, Kt/V and baseline values of 6MWT, the type of training remained significantly associated with the amount of increase in walked distance.

Although the best protocol of exercise for patients on dialysis is not yet clear, in the investigators sample of hemodialysis patients the combination of aerobic and resistance training was more effective to improve functional performance.

ELIGIBILITY:
Inclusion Criteria:

* to be on hemodialysis therapy for longer than 3 months
* to be already included in the resistance training protocol during dialysis
* to receive erythropoietin for the treatment of anemia
* hemoglobin level greater than 9.0 g/dL
* to be able to maintain sitting and standing balance and ambulatory without assistance.

Exclusion Criteria:

* symptomatic ischemic heart disease
* recent myocardial infarction of less than 6 months
* uncontrolled hypertension
* pericardial or pleural friction rub
* aortic stenosis
* active musculoskeletal lower-extremity problem, or history of vertebral fracture caused by osteoporosis
* patients were also excluded if they participated in formal organized exercise programs outside the dialysis unit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
physical performance | 10 weeks

SECONDARY OUTCOMES:
dialysis adequacy (KtV) | 4/8/10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitário São Francisco de Paula, Pelotas, Rio Grande do Sul, Brazil